CLINICAL TRIAL: NCT04885699
Title: Validation of Capnodynamic Assessment of Mixed Venous Oxygen Saturation and Cardiac Output in Anesthetized Children Undergoing Cardiac Catheterization
Brief Title: Validation of Capnodynamic Assessment of Mixed Venous Oxygen Saturation
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Jacob Karlsson, Principal Investigator, Karolinska Institutet
Other Study IDs: KarolinskaALB
Record Dates: First submitted 2021-05-09; First posted 2021-05-13 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2024-10

CONDITIONS: Cardiac Output, Low; Cardiac Output, High
Keywords: mixed venous oxygen saturation; capnodynamics
MeSH Terms: conditions — Cardiac Output, Low; Cardiac Output, High

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Mixed venous saturation (SvO2) is an indicator of the balance between oxygen supply and demand in the body's tissues Recently, our research team published a paper describing the possibility to continuously monitor SvO2 by the use of continuous dynamic capnography (Karlsson et al, A Continuous Noninvasive Method to Assess Mixed Venous Oxygen Saturation: A Proof-of-Concept Study in Pigs. Anesth Analg 2020) The primary objective of the current study is thus to investigate the agreement and trending ability for capnodynamically derived SvO2 against the gold standard CO-oximetry. The secondary objective is to investigate the agreement and trending ability for capnodynamically derived CO (COEPBF) against the modified CO2-Fick method.

DETAILED DESCRIPTION:
Background: Mixed venous saturation (SvO2) is an indicator of the balance between oxygen supply and demand in the body's tissues The primary objective of the current study is thus to investigate the agreement and trending ability for capnodynamically derived SvO2 against the gold standard CO-oximetry. The secondary objective is to investigate the agreement and trending ability for capnodynamically derived CO (COEPBF) against the modified CO2-Fick method.

Methods:

The rationale of capnodynamic SvO2 (capno-SvO2) can be briefly described as follows:

The Capno-SvO2 method is based on differential Fick's principle and utilizes a combination of continuous estimation of Effective Pulmonary Blood Flow (COEPBF) and oxygen consumption (VO2) incorporated in a rearranged Fick's equation. COEPBF is estimated by applying a special breathing pattern of variations in I:E relationships (six breaths with normal I:E relations followed by three breaths vid an approximately 2 s expiratory pause). This breathing pattern causes small fluctuations in alveolar CO2 concentration and VCO2, related to the pulmonary blood flow participating in gas exchange which allows for estimation of COEPBF. VO2 can be estimated using continuous volumetric capnography measurement of VCO2 combined with the Respiratory Quotient (RQ).

Modified CO2-Fick: CO estimation using modified CO2-Fick is assessed by incorporating measured CO2 content in mixed venous and arterial blood into the equation below where VCO2 is estimated using volumetric capnography.

COFick=VCO2/(CvCO2-CcCO2)

Study protocol

All patients planned for percutaneous intervention of cardiac conditions at our department will be screened for inclusion in this study. Exclusion criteria: ongoing ECMO treatment or intracardiac shunts not subjected to intervention. All these patients are routinely anaesthetized, intubated with a cuffed endotracheal tube and kept on controlled ventilation, a prerequisite for the capnodynamic method.

After induction of anesthesia, the special breathing pattern will be applied and continuous data from the capnodynamic monitoring will be collected. After catheterization of the pulmonary artery two baseline blood gases from the PAC and arterial line will be drawn and analyzed, and the hemoglobin level (Hb) from this sample will be used for calibration of the capnodynamic method together with a tabulated RQ. After completion of the interventional procedure, a sequence of paired testing of SvO2 from blood gases drawn from the pulmonary artery and arterial line. Firstly 2 samples (3 min apart) forming a baseline. After this follows a short increase in PEEP (3 cmH2O to 8cmH2O), which temporarily decreases cardiac output and SvO2. A sample is collected and then once more after PEEP has been brought back to 3 cmH2O after 3 minutes. Next, a raised level of inhaled oxygen from 30 to 80% (FiO2) is applied for 3 minutes and then turned back to baseline. Mixed venous and arterial samples will be drawn at FiO2 30% and 80%.

Paired recordings of COEPBF and CO2-Fick as well as capnodynamic SvO2 and co-oximetry will be examined for agreement and ability to detect change using Bland-Altman and four quadrant plots.

Power analyses (power 80% and alfa of 0.05) implies a minimal of 120 paired recordings corresponding to approximately 20 patients. 30 patients will be included for upward margin.

ELIGIBILITY:
Inclusion Criteria: Patients undergoing percutaneous intervention of cardiac conditions such as closure of atrial septal defect, persistent ductus arteriosus, pulmonary artery stenosis and diagnostic catheterization after heart transplant.

-

Exclusion Criteria: ongoing ECMO treatment or intracardiac shunts not subjected to intervention. Weight less than 3.5 kg. Single ventricle circulation.

-

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Full term newborn children up till 18 years of age undergoing interventional/diagnostic cardiac catheterization
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Capnodynamic Mixed venous oxygen saturation vs CO-oximetry | 20 minutes
  Agreement of absolute values between Capnodynamic Mixed venous oxygen saturation and the reference method CO-oximetry

SECONDARY OUTCOMES:
Agreement of absolute values between Capnodynamic cardiac output and the reference method modified CO2-Fick | 20 minutes
  Comparing continuous capnodynamic measurement of effective pulmonary blood flow (cardiac output) and CO obtained by modified CO2-Fick.

CONTACTS AND LOCATIONS:
Overall Officials: Per-Arne Lönnqvist, MD, Study Chair — Karolinska University
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No